CLINICAL TRIAL: NCT06916572
Title: Effects of Scapular Stabilization Exercises and Scapular Proprioceptive Neuromuscular Facilitation Technique on Pain, Range of Motion, Functionality, Scapular Dyskinesia and Proprioception in Patients With Rotator Cuff Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Zeynep HOŞBAY, Professor, Physiotherapist, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Scapula in rotator cuff lesion
Record Dates: First submitted 2025-03-12; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff Lesions
Keywords: Rotator Manşet Lezyonu; Skapular PNF Tekniği; Propriosepsiyon; Skapular Stabilizasyon Egzersizi; Skapula

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial
Who Masked: Participant
Masking Description: Participants does not know which type of treatment is received themselves.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Scapular Stabilization Group (Experimental): The scapular stabilization exercises applied in addition to conventional treatment are as follows:
  Clock Exercise on the Wall Dynamic Stabilization Exercises on the Wall Push-Up Exercise on the Wall Retraction Exercises Scapular Depression Exercise Double Arm Balance Exercise
  Interventions: Other: Scapular stabilization exercises
- PNF Group (Experimental): The scapular PNF patterns of anterior elevation - posterior depression and anterior depression - posterior elevation were applied with rhythmic initiation, repeated contractions (stretches) and rhythmic stabilization techniques with 10 repetitions of each technique.
  Interventions: Other: Scapular PNF

INTERVENTIONS:
Other: Scapular stabilization exercises — Individuals in the Scapular Stabilization group received a physiotherapy and rehabilitation program for 6 weeks, 3 days a week. The treatment of individuals in this group included scapular stabilization exercises in addition to conventional treatment. Scapular stabilization exercises were planned to be applied only on the days of the session. Each of the exercises was applied as 10 repetitions and 2 sets.
  Conventional treatment included an exercise program consisting of Wand, Codman, finger ladder and rotator cuff strengthening exercises, in addition to 20 min HotPack, 20 min TENS and 5 min Ultrasound modalities.
  Arms: Scapular Stabilization Group
Other: Scapular PNF — Physiotherapy and rehabilitation program was applied to the individuals in the PNF group for 6 weeks, 3 days a week, as in the Scapular Stabilization group. In addition to conventional treatment, scapular PNF approaches were added to the treatment of individuals in this group.
  The scapular PNF patterns of anterior elevation - posterior depression and anterior depression - posterior elevation were applied with rhythmic initiation, repeated contractions (stretches) and rhythmic stabilization techniques with 10 repetitions of each technique.
  Conventional treatment included an exercise program consisting of Wand, Codman, finger ladder and rotator cuff strengthening exercises, in addition to 20 min HotPack, 20 min TENS and 5 min Ultrasound modalities.
  Arms: PNF Group

SUMMARY:
This study aimed to compare the effects of Scapular Proprioceptive Neuromuscular Facilitation (PNF) applications and Scapular Stabilization exercises on pain, joint range of motion, functionality, scapular dyskinesia, and proprioception in individuals with rotator cuff lesions. The study included 30 volunteer participants aged 18 to 65 years, who had been diagnosed with Rotator Cuff Lesion and reported shoulder pain. The Scapular Stabilization group (n=15) received scapular stabilization exercises in addition to conventional treatment, while the PNF group (n=15) received scapular PNF patterns and techniques in addition to conventional treatment. In this study, the Visual Analog Scale (VAS) was used to evaluate the pain severity of individuals, a universal goniometer was used to measure joint range of motion, and the Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) was used to assess functional status. Scapular dyskinesia was evaluated using the Lateral Scapular Shift Test (LSKT) and Scapular Dyskinesia Test (SDT), while proprioception was assessed using the Active Angle Repetition Test. Statistical analysis of the data was performed using SPSS V.27 software.

DETAILED DESCRIPTION:
The shoulder joint, also known as the glenohumeral joint, is a dynamic structure that can move in the sagittal, vertical and transverse planes, offering the widest range of motion in the human body. The humeral head articulates with the glenoid fossa of the scapula to form the glenohumeral joint, which is the main joint of the shoulder girdle. The glenohumeral system allows movement in multiple axes thanks to static and dynamic stabilizing structures, but the flexibility of these structures increases the risk of shoulder instability. The scapula is a triangular-shaped bone that supports shoulder functions, which are the cause of anatomy and biomechanical properties; It acts as a platform to which the muscles are attached, connecting the glenohumeral joints to the body and the glenohumeral joints. In a healthy shoulder girdle, the scapula should provide a stable base and the scapular muscles should provide a dynamic position during shoulder joint movements.

Rotator cuff muscles are an important muscle group that plays a role in scapular stabilization by coordinating this dynamic balance with glenohumeral extension strength and is a training aid for scapulohumeral rhythm. Weakness or dysfunction in the scapular muscles disrupts the scapulohumeral rhythm and becomes open to sports in the glenohumeral regions, which play an important role in daily living activities (ADL). The most common degenerative sports seen around the glenohumeral joints are Rotator Cuff Lesions and those that can be found completely or partially according to the parts of the lesions. The risk of occurrence continues to increase with age; It is seen at a rate of 4% in individuals aged 40 and over, while it is seen at a rate of 54% in individuals aged 60 and over. Individuals with rotator cuff pain in the shoulder, the range of motion in between, and the average duration are observed as if they were not impaired. In cuff lesions, the function of the structures responsible for the stabilization of the scapula cannot be performed due to the decrease in the biomechanics of the scapula and the functionality is negatively affected. Rotator cuff lesions can be treated with conservative or surgical intervention. The age of the patient, general health status, aging of the lesion and its functioning are the completion of the treatment accumulation of parts. In cuff lesions, conservative cuts such as medical treatment and physiotherapy applications are usually preferred first, but surgical interventions can be resorted to in cases where this treatment is insufficient. Conservative management of rotator cuff lesions, additional range of motion exercises, stretching and strengthening routines, manual therapy techniques, hot-cold applications or different treatment methods such as transcutaneous electrical nerve stimulation (TENS) can be used. Scapular stabilization exercises are a group of exercises that support shoulder functions and ensure continuity of scapular movement by ensuring that the scapula and humerus work in harmony. This group of exercises should be added to the treatment to regulate the scapulohumeral rhythm affected by rotator cuff lesions and to reactivate normal shoulder capacity. Proprioceptive neuromuscular facilitation (PNF) treatments, which help facilitate neuromuscular mechanism responses by stimulating proprioceptors, are also planned as a treatment approach for neuromuscular treatment of the scapula with the inclusion of conservative treatment methods.

There are studies in the literature on shoulder PNF pattern and techniques and scapular stabilization exercises in individual parts with rotator cuff lesions. However, it has been observed that the treatment of scapular PNF pattern and techniques and scapular stabilization exercises and the symptoms comparing the effectiveness of these two treatment approaches on the effect are not sufficient.

The purpose of this process is to compare whether the scapular stabilization exercises and scapular PNF pattern and techniques on the sound, range of motion of the joints, functionality, scapular dyskinesia and proprioception in individuals with rotator cuff parts and the support of these two treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 - 65 years of age
* Getting a diagnosis of Rotator Cuff Lesion,
* Presence of unilateral shoulder pain for a minimum of 3 weeks,
* Signing the "Informed Voluntary Consent Form",
* Individuals who are cooperative and willing to participate in the study.

Exclusion Criteria:

* Corticosteroid treatment or local corticosteroid injections in the last three months,
* Neer Stage 3 tear of the rotator cuff tendons,
* Shoulder fracture or instability,
* Physiotherapy within the last 6 months on the same shoulder,
* History of surgery in the shoulder girdle or thorax,
* With cognitive and mental problems,
* Individuals with malignancy, neuromuscular disorders, unstable angina, arthritis, cardiopulmonary disorders, vertigo or various vestibular system disorders and communication problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain | 6 weeks
  In our study, pain was assessed using the Visual Analog Scale (VAS). The Visual Analog Scale is a scale in which pain intensity is expressed by marking on a line 0-10 cm long. Before the assessment, participants were informed that the numbers on the scale were expressed as "'0: no pain' and '10: unbearable pain'" and were asked to mark the intensity of pain they felt at rest, during activity, and at night on the line.
Range of Motion of the Shoulder Joint | 6 weeks
  In our study, individuals' shoulder joint range of motion was measured with a "universal goniometer" and evaluated. Goniometric measurement is an objective method frequently used in ROM evaluation. Before and after treatment, individuals' shoulder flexion, extension, abduction, external rotation and internal rotation active and passive range of motion was measured with a universal goniometer. Measurements were made 3 times and the average of each measurement was recorded.
Shoulder Functionality | 6 weeks
  In the study, the Turkish translated version of the Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH), which consists of three sections, was used to assess the functional limitation and disability status of the upper extremity. The first part (DASH-FS) includes 30 questions to assess the individual's limitations in activities of daily living, symptoms experienced and functional status in social life. The second section (DASH-W) is related to the work model. This section inquires about the patient's limitations and disability status in working life. The third section (DASH-SM) assesses the functional limitations of those who are professionally involved in music or sports. For each question of the questionnaire, a 5-point Likert response scale (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: no difficulty at all) is used. The patient gives the appropriate response and a total score between 0-100 is obtained.
Scapular Dyskinesia | 6 weeks
  The "Scapular Dyskinesia Test (SDT)" was used to evaluate the dynamic movement of the scapula. During the test, the patient was asked to perform bilateral full shoulder elevation with the elbow in extension and shoulder in neutral position with weights determined on the basis of his/her current weight in the standing position and to slowly lower his/her arms when he/she reached the final degree. During the test, individuals with a body weight of 68.1 kg and above were asked to complete the maneuver using a dumbbell weighing 2.3 kg, and individuals with a body weight of less than 68.1 kg were asked to complete the maneuver using a dumbbell weighing 1.4 kg. The test was repeated 3 times. Scapular movements during the test maneuver were evaluated observationally. The type of dyskinesia was determined according to "Kibler's Scapular Dyskinesia Evaluation System" and the observed asymmetry was recorded.
Scapular Dyskinesia | 6 weeks
  The lateral scapular shear test (LSST) is a static test based on bilateral measurement of the distance between the inferior end of the scapula and the processus spinosus of the aligned vertebra. The measurement was performed in 3 different positions in standing posture; arms at the side of the trunk in the resting position, hands on the waist, shoulder in 45º abduction position and shoulder in maximum internal rotation and 90º abduction position. Measurements were made with a tape measure and the results were recorded in "cm". In these three positions, scapular dyskinesia was recorded as positive when the distance difference between the two sides was 1.5 cm or more.
Shoulder Proprioception | 6 weeks
  In our study, shoulder joint proprioception was evaluated using the "active angle repetition test". During the test, position sense was considered normal in individuals whose absolute value of the difference between the determined angle and the angle reached by the patient was below 6.6°, while position sense was considered lost in individuals whose absolute value was 6.6° and above. Active angle repetition test was performed using a target board and laser pointer. Individuals were asked to perform a 40° shoulder elevation with their eyes open and repeat this three times. Then, individuals were asked to close their eyes to eliminate visual sensory support and find the target angle they learned. This process was repeated 6 times. The same test was applied for another target angle, 100°. The same process was repeated for each trial and the averages were calculated and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin YL, Karduna A. Exercises focusing on rotator cuff and scapular muscles do not improve shoulder joint position sense in healthy subjects. Hum Mov Sci. 2016 Oct;49:248-57. doi: 10.1016/j.humov.2016.06.016. Epub 2016 Jul 29. PMID 27475714
- [Background] Bakhsh W, Nicandri G. Anatomy and Physical Examination of the Shoulder. Sports Med Arthrosc Rev. 2018 Sep;26(3):e10-e22. doi: 10.1097/JSA.0000000000000202. PMID 30059442